CLINICAL TRIAL: NCT01369264
Title: Evaluation of the Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Brain Electrical Activity in Healthy Human Volunteers
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation on Brain Activity in Healthy Human Volunteers
Acronym: ERP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Gary M. Hasey, MSc, MD, FRCPC, McMaster University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 07-2827
Record Dates: First submitted 2010-09-18; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2007-07

CONDITIONS: Changes in EEG During and After Magnetic Stimulation
Keywords: Repetitive Transcranial Magnetic Stimulation (rTMS); Electroencephalography (EEG); Magnetic Resonance Imaging; Quantitative EEG (QEEG)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- True Left High Frequency (Experimental): True left high frequency repetitive transcranial magnetic stimulation
  Interventions: Device: true left high frequency
- Passive sham left high frequency (Placebo Comparator): Passive sham left high frequency repetitive transcranial magnetic stimulation
  Interventions: Device: Passive sham left high frequency

INTERVENTIONS:
Device: true left high frequency — 10 Hz stimulation will be given at 110% motor threshold for 8 seconds to Brodmann areas 46, 9 and 10 in the left hemisphere. The coil will be held flat over the skull surface with the coil handle held at approximately 45 degrees to the floor
  Other Names: Magstim super rapid left true 10 Hz
  Arms: True Left High Frequency
Device: Passive sham left high frequency — 10 Hz stimulation will be given at 110% motor threshold for 8 seconds to Brodmann areas 46, 9 and 10 in the left hemisphere. The passive (inactive) coil will be held flat over the skull surface with the coil handle held at approximately 45 degrees to the floor. An active coil will be held vertically in a mechanical holder 50 cm behind the subject head and run at 10 Hz with an intensity set to 150% of motor threshold.
  Other Names: Magstim super rapid left passive sham 10 Hz
  Arms: Passive sham left high frequency

SUMMARY:
The proposed study is designed to determine whether small changes in the positioning of a transcranial magnetic stimulation coil over the frontal parts of the brain cause different patterns of brain activation measured by electroencephalography (EEG) and quantitative EEG (QEEG).

DETAILED DESCRIPTION:
A previously recorded MRI will be loaded into Brainsight, a stereotactic neuronavigation system specifically designed to be used with rTMS, and the scalp surface site overlying the centre of Brodmann area 46 in the dorsolateral prefrontal cortex (DLPFC) of both the left and right hemisphere will be identified and marked on a spandex swim cap placed on the subjects head over 31 EEG electrodes (notched to prevent eddy currents) placed at international 10-20 locations . Three trains of true 10 Hz (110% motor threshold (MT)] rTMS (one train each with duration=2,4, and 8 seconds) and 6 similar trains of sham rTMS (3 of active sham and 3 of inactive sham) will be delivered to the left hemisphere in Brodmann area 46 in random order. Eyes-closed QEEG power will be recorded across all leads over 10 second "blocks" for 1 minute after each 10 Hz stimulus to determine the distribution and time course of any changes in electrical potential and QEEG spectrum. The subjects will be asked to rate their mood and anxiety by placing a mark along 100 mm long Visual Analogue Scales for depression and anxiety after each stimulus train. We will also measure ERPs after 1 Hz stimulation to the right DLPFC (centre of Brodmann area 46). We will administer three 60-second trains of true 1 Hz rTMS (at 90%, 100% and 110% motor threshold), and six 60-second trains of sham rTMS (3 of "active" sham and 3 of "inactive" sham) with device intensity setting of 10 %, 30% and 50% motor threshold and coil tilted at 90 degrees away form the head. Part 2 (location testing): Twenty four to 48 hours later, the swim hat will be placed on the subject's head and the neuroanatomical landmarks reconfirmed using Brainsight. One true train and 1 inactive sham train of 10 Hz rTMS (10 Hz, 110% MT) will be delivered in random order to Brodmann area 46 and two other sites (in Brodmann areas 9 and 10). The rTMS train duration will be 8 seconds. The subjects will be asked to rate their mood and anxiety by placing a mark along 100 mm long Visual Analogue Scales for depression and anxiety after each stimulus train. The same procedure will be done over the right hemisphere using 1 Hz stimulation set at 110% motor threshold. True rTMS pulses at 1 Hz, or inactive sham rTMS pulses will be delivered in 60 second trains to the 3 sites as described above, but marked over the right DLPFC. QEEG activity will be recorded for 1 minute after each stimulus train. The subjects will be asked to rate their mood and anxiety by placing a mark along 100 mm long Visual Analogue Scales for depression and anxiety after each stimulus train. Diffusion Tensor Imaging: The 15 healthy subjects (18-65 years old) will also undergo diffusion tensor imaging (DTI) along with the MRI, which will add approximately 10 minutes to the MRI procedure. Following a routine brain imaging protocol whole brain DTI measurements will be conducted in each subject using a single shot spin echo EPI diffusion tensor imaging sequence.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* male or female

Exclusion Criteria:

* uncontrolled physical health problems
* psychiatric illness
* personal and/or family history of epilepsy/seizures
* metal in the head or neck
* recent head injury
* pacemaker
* pregnancy
* alcohol/substance abuse within 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be global mean field amplitude (GMFA) before and after treatment with true or sham rTMS using a range of stimulus train durations and several stimulation sites. | The GMFA will be measured for 1 minutes after each rTMS train is delivered.

SECONDARY OUTCOMES:
Secondary outcome measures will include magnetically evoked response potentials in the multi-channel recorded EEG signals. | The L/R APR will be measured for 1 minute after each TMS train is delivered.
  The magnetically evoked response potentials will be measured over the first 500 milliseconds after each TMS pulse.
  We will also determine weather rTMS can produce measurable changes in left/right alpha power ratio (L/R APR). The L/R APR will be measured for 1 minute after each TMS train is delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hasey, MD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Healthcare, Centre for Mountain Health Services, Hamilton, Ontario, Canada